CLINICAL TRIAL: NCT01701206
Title: Using Online Social Networks for HIV Prevention and Testing
Brief Title: HOPE (Harnessing Online Peer Education): Using Online Social Networks for HIV Prevention and Testing
Acronym: HOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Sean Young, PhD, MS, Assistant Professor In-Residence, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: K01MH090884 (NIH)
Record Dates: First submitted 2012-10-04; First posted 2012-10-05 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: HIV
Keywords: HIV; social networking; at-risk populations; sexual risk behaviors

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- HIV intervention Group (Experimental): Experimental arm receives peer-led HIV information on social media
  Interventions: Behavioral: HIV knowledge Intervention
- Control arm (No Intervention)

INTERVENTIONS:
Behavioral: HIV knowledge Intervention
  Arms: HIV intervention Group

SUMMARY:
This study seeks to determine whether social networking technologies can be used to increase HIV prevention and testing.The HOPE (Harnessing Online Peer Education) model seeks to apply a diffusion of innovations style intervention to social media to increase HIV testing.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Has had sex with a man in the past 12 months
* Lives in Lima or Callao, Peu
* Has a Facebook account or willing to create one

Exclusion Criteria:

* Does not satisfy inclusion criteria

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2009-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
HIV self-testing-Number of participants who request an HIV self-testing kit | Measured during the intervention

CONTACTS AND LOCATIONS:
Locations (2):
- University of California, Los Angeles, Los Angeles, California, United States
- Epicentro Commun, Lima, Peru

REFERENCES:
- [Derived] Young SD, Cumberland WG, Nianogo R, Menacho LA, Galea JT, Coates T. The HOPE social media intervention for global HIV prevention in Peru: a cluster randomised controlled trial. Lancet HIV. 2015 Jan;2(1):e27-32. doi: 10.1016/S2352-3018(14)00006-X. PMID 26236767
- [Derived] Young SD, Cumberland WG, Lee SJ, Jaganath D, Szekeres G, Coates T. Social networking technologies as an emerging tool for HIV prevention: a cluster randomized trial. Ann Intern Med. 2013 Sep 3;159(5):318-24. doi: 10.7326/0003-4819-159-5-201309030-00005. PMID 24026317